CLINICAL TRIAL: NCT00112060
Title: A Phase I/II, Open-Label, Multicenter Study of Single Agent PT-523 in the Treatment of Relapsed or Refractory Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study to Assess the Safety and Preliminary Efficacy of PT-523 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBS101; HBS101.00
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Talotrexin; PT-523; Non-Small Cell Lung Carcinoma (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — N(alpha)-(4-amino-4-deoxypteroyl)-N(delta)-hemiphthaloyl-L-ornithine; Injections

INTERVENTIONS:
Drug: PT-523 for Injection

SUMMARY:
This phase I/II, multi-centered, non-randomized trial is designed to determine a safe dose of PT-523 for subjects, and to make preliminary evaluations on the activity of PT-523 as therapy in subjects with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed NSCLC which is stage III or stage IV, or recurrent disease, and failed therapy with a standard first line (Phase I/II) as well as second line chemotherapy regimen (Phase I), or be intolerant of standard chemotherapy. Receipt of one additional prior chemotherapy regimen for neoadjuvant, adjuvant, or neoadjuvant plus adjuvant is allowable. A prior epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TK) antagonist is allowable (Phase II).
* Asymptomatic or treated brain metastases (including steroids) if last therapy was received > 4 weeks from study entry and is deemed by the investigator to have a low likelihood of rapid deterioration.
* ECOG performance status 0 - 2.
* Adequate organ function and bone marrow reserve.
* Use of appropriate contraceptive method.
* Signed patient informed consent.

Exclusion Criteria:

* Investigational agents within 30 days prior to Day 1 of study.
* Known symptomatic or uncontrolled brain metastases.
* Uncontrolled intercurrent illness.
* Known human immunodeficiency virus (HIV), hepatitis A, B, C, D and E.
* Patient has uncontrolled pleural effusions.
* Patient has received nitrosoureas or mitomycin-C within 6 weeks or other chemotherapy or radiation therapy within 3 weeks before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - University of Miami and Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University & University Hospitals of Cleveland, Cleveland, Ohio
- Russia (9):
  - Chelyabinsk Regional Oncology Center Chemotherapy Department, Chelyabinsk
  - Irkutsk Regional Oncology Center, Irkutsk
  - Blokhin Cancer Research Center Department of Chemotherapy and Combination Treatment of Neoplasia, Moscow
  - Blokhin Cancer Research Center Department of Clinical Pharmacology and Chemotherapy, Moscow
  - Semashko Central Clinical Hospital, Moscow
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Petrov Research Institute of Oncology, Saint Petersburg
  - St. Petersburg Oncology Center Thoracic Department, Saint Petersburg
  - Yaroslavl City Oncology Center, Yaroslavl

REFERENCES:
- See also: Hana Biosciences, Inc. is a South San Francisco, CA - based biopharmaceutical company that acquires, develops, and commercializes innovative products to advance cancer care. — http://www.hanabiosciences.com